CLINICAL TRIAL: NCT04583930
Title: Clinical and Health-related Outcome of rFVIIIFc Prophylaxis in Patients With Haemophilia A
Brief Title: Clinical and Health-related Outcome of rFVIIIFc Prophylaxis
Acronym: CLHEAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Dr. Dr. Thomas Hilberg (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dr. Thomas Hilberg, Head of Department, University of Wuppertal
Organization: University of Wuppertal (Other)
Other Study IDs: Hae-Ger-2019-251-Hil
Record Dates: First submitted 2020-07-28; First posted 2020-10-12 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Haemophilia A: * Patients suffering from moderate to severe haemophilia A
  * Age ≥ 18-years
  * Treatment with FVIII prophylaxis
  * Submitted written informed consent

SUMMARY:
Current standard therapy for patients with haemophilia (PwH) in the prevention of bleeding episodes is a prophylactic intravenous treatment with recombinant coagulation factor (F) VIII (Haemophilia A) or rather FIX (Haemophilia B) two to three times weekly. With the development of recombinant factor VIII Fc fusion protein (rFVIIIFc) the conventional routine prophylaxis regime is complemented by an extended half-life (EHL) factor replacement prophylaxis with the potential of improved bleed prevention and reduced injection frequency at similar factor consumption. Aim of this longitudinal multicentre study is to evaluate the influence of an EHL factor replacement regime with rFVIIIFc on haemophilic specific parameters (annual bleeding rate, bleeding localisation), joint status, pain, functional parameters, treatment adherence and health-related quality of life in PwH A.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from moderate to severe haemophilia A
* Age ≥ 18-years
* Treatment with FVIII prophylaxis
* Submitted written informed consent

Exclusion Criteria:

Patients suffering from other bleeding diseases

* Patients with inhibitors
* Patients without written informed consent
* Age < 18-year-old
* Any surgeries up to 6 months before the examination date
* Suffering from different rheumatologic diseases like M. Bechterew, Psoriasis or other local or generalized joint infections (Borreliosis, septic arthritis)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate or severe Haemophilia A will be included in this study consecutively, who will be switched from FVIII prophylaxis on rFVIIIFc prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
total annual bleeding rate | one year
  number of total bleedings
orthopaedic joint status (Haemophilia health joint score) | one year
  The clinical joint status will be examined in all patients with haemophilia by the World Federation Joint Examination Score and Haemophilia Joint Health Score. Higher score points imply an increased deficit in the functional and structural joint status as a sign of more pronounced haemophilic arthropathy, with a maximum possible value of 124 (no deficits = 0).
pressure pain thresholds | one year
  physiological Parameter in Newton

SECONDARY OUTCOMES:
spontaneous joint ABR | one year
  number of total joint bleedings
subjective quality of life (SF-36) | two years
  The standarized questionnaire SF-36 includes a physical and psychological score. The higher the score, the higher the physical or psychological quality of life. A higher score implies a better physical and mental quality of life
subjective physical performance (HEP-Test-Q) | two years
  The final version of the standarized questionnaire consists of 25 items pertaining to the domains 'mobility', 'strength & coordination', 'endurance' and 'body perception'. The response options were a five-point Likert scale (ranging from 1 = never to 5 = always). Some of the items had to be re-coded; subscales and the total score were transformed to a scale of 0-100 with high scores indicating better physical performance
self-perceived functional abilities (Haemophilia Activities List) | two years
  The Haemophilia Activities List measures the impact of hemophilia on self-perceived functional abilities in adults. It contains 42 multiple choice questions in seven domains: Lying/sitting/kneeling/standing (8 items), Functions of the legs (9 items), Functions of the arms (4 items), Use of transportation (3 items), Self-care (5 items), Household tasks (6 items), Leisure activities and sports (7 items)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hilberg, Prof., Principal Investigator — Head of Department
Locations (2):
- Germany (2):
  - Department of Sports Medicine, University of Wuppertal, Wuppertal, North Rhine-Westphalia
  - Department of Sports Medicine, Wuppertal, Northwest

IPD SHARING:
Plan to Share IPD: No